CLINICAL TRIAL: NCT00207844
Title: Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating Efficacy and Safety of a Therapeutic Administration of Selenium, as Selenite, in Septic Shock Patients.
Brief Title: Selenium, as Sodium Selenite, in the Treatment of Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier de Meaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFSSAPS 10602; CIC0203/003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Selenium; Oxidative stress; Septic shock; Sodium selenite
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Selenium; Sodium Selenite

INTERVENTIONS:
Drug: Selenium as sodium selenite

SUMMARY:
Septic shock is a frequent syndrome with a 45% mortality rate despite intensive care unit (ICU) care, where free radicals may play a key role, and a >40% decrease in plasma selenium concentration is observed. Selenium is a trace element with both indirect enzymatic anti-oxidant, and direct oxidant properties. High dose of sodium selenite administration could increase antioxidant cells capacities, and reduce inflammation by a direct paradoxical pro-oxidative effect. We conduct a study to evaluate the effects of selenium treatment in comparison to placebo, in septic shock patients. Efficacy will be evaluated by the weaning time of catecholamines.

DETAILED DESCRIPTION:
Septic shock - an uncontrolled systemic host response to invasive infection -, leading to multiple organ failure, is a public health issue because of its frequency (> 1/1000 inhabitants per year), its cost and its 45% mortality rate, remaining high despite all the improvements made in ICU for the past 20 years. His physiopathology is better understood with increasing data supporting the key role of free radicals, and a more than 40% plasma selenium concentration decrease that maybe associated with increased morbidity and mortality. Meanwhile, for the past 30 years, researches have been conducted on the essential trace element selenium for its requirement for key antioxidant enzymes, through the 21st aa selenocystein, and also for its potentially toxic, pro-oxidant properties. In septic shock, both properties may be useful, antioxidant enzymatic to increase cell defense especially endothelial cells, and direct pro-oxidant action to decrease the genomic response, especially on phagocytic cells.

The objective of this study is to evaluate the effects of a high dose of selenium administration, such as selenite, at pro-oxydant initial dose followed by anti-oxidant dose in severe septic shock patients with documented infection. The initial dose was chosen as the highest dose of selenium, as sodium selenite, estimated without severe adverse effects in healthy people for a one-day ingestion. The patients are randomized to receive either the placebo or the selenite at this high initial dose followed by lower doses on a 9-day period. The efficacy will be evaluated by the weaning time of catecholamines, with a special attention to the 6-month mortality rate as first secondary end point.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in ICU
* Severe documented infection
* Ventilation
* Circulatory failure requiring high dose of catecholamine
* IGS II score >25 at inclusion
* Informed written consent

Exclusion Criteria:

* Pregnancy
* End phase chronic disease
* Limitation of care
* Shock due to an urinary infection without bacteriemia
* Peritonitis related to peritoneal dialysis or trauma
* Preliminary circulatory failure
* Participating to another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-01; Study Completion 2005-01

PRIMARY OUTCOMES:
Weaning time of catecholamines

SECONDARY OUTCOMES:
- 6 month mortality rate
- 6 month quality of life
- 28 days mortality
- ICU mortality
- Hospital mortality
- ICU length of stay
- Hospital length of stay
- Number of nosocomial infections in ICU
- Duration of ventilation
- SOFA score in ICU at days 4, 7, 10 and 14
- Oxidative stress evaluation at days 4, 7, 10 and 14
- Inflammation evaluation at days 4, 7, 10 and 14
- Selenium status
- Costs and work load
- Onset of clinical events

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Forceville, MD, Principal Investigator — CH Meaux; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (7):
- France (7):
  - Service de Réanimation - Centre Hospitalier Victor Dupouy, Argenteuil
  - Service de Réanimation Polyvalente - CH de Châlons, Châlons-en-Champagne
  - Service de Réanimation Médicale - Hôpital Raymond Poincaré, Garches
  - Service de Réanimation - HIA Desgenettes, Lyon
  - Service de Réanimation Polyvalente - Hôpital Saint Faron, Meaux
  - Service Réanimation - HIA Saint Anne, Toulon
  - Service de Réanimation - Centre Hospitalier G. Dron, Tourcoing

REFERENCES:
- [Background] Brun-Buisson C, Doyon F, Carlet J, Dellamonica P, Gouin F, Lepoutre A, Mercier JC, Offenstadt G, Regnier B. Incidence, risk factors, and outcome of severe sepsis and septic shock in adults. A multicenter prospective study in intensive care units. French ICU Group for Severe Sepsis. JAMA. 1995 Sep 27;274(12):968-74. PMID 7674528
- [Background] Forceville X, Vitoux D, Gauzit R, Combes A, Lahilaire P, Chappuis P. Selenium, systemic immune response syndrome, sepsis, and outcome in critically ill patients. Crit Care Med. 1998 Sep;26(9):1536-44. doi: 10.1097/00003246-199809000-00021. PMID 9751590
- [Background] Goode HF, Webster NR. Free radicals and antioxidants in sepsis. Crit Care Med. 1993 Nov;21(11):1770-6. doi: 10.1097/00003246-199311000-00029. PMID 8222696
- [Background] Novelli GP. Role of free radicals in septic shock. J Physiol Pharmacol. 1997 Dec;48(4):517-27. PMID 9444605
- [Derived] Forceville X, Laviolle B, Annane D, Vitoux D, Bleichner G, Korach JM, Cantais E, Georges H, Soubirou JL, Combes A, Bellissant E. Effects of high doses of selenium, as sodium selenite, in septic shock: a placebo-controlled, randomized, double-blind, phase II study. Crit Care. 2007;11(4):R73. doi: 10.1186/cc5960. PMID 17617901